CLINICAL TRIAL: NCT01985230
Title: Investigation of the ReActiv8 Implantable Stimulation System for Chronic Low Back Pain
Brief Title: ReActiv8 for Chronic Low Back Pain (PMCF)
Acronym: ReActiv8-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mainstay Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 950002
Record Dates: First submitted 2013-11-05; First posted 2013-11-15 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ReActiv8 Implant (Experimental)
  Interventions: Device: ReActiv8 Implantable Stimulation System implanted and activated.

INTERVENTIONS:
Device: ReActiv8 Implantable Stimulation System implanted and activated.

SUMMARY:
The purpose of this Clinical Study is to investigate the effect of electrical stimulation for chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, ≤65 years
2. Chronic Low Back Pain with a first occurrence >90 days prior to enrolment, and the last relatively pain-free time >90 days prior to enrolment.
3. Continuing low back pain despite >90 days of medical management
4. Oswestry Disability Index score ≥25% and ≤60% at the time of enrolment
5. Able to understand and sign the Informed Consent form.
6. Ability to comply with the instructions for use and to operate the ReActiv8, and to comply with this Clinical Investigation Plan.
7. Suitable for ReActiv8 surgery as determined by the implanting physician prior to inclusion.
8. Prior week average Low Back Pain NRS of ≥6.0 and ≤9.0 on a 11 point NRS scale (0-10) at the Baseline Visit

Exclusion Criteria:

1. BMI > 35
2. Back Pain characteristics:

   1. Any surgical correction procedure for scoliosis at any time, or a current clinical diagnosis of scoliosis.
   2. Lumbar spine stenosis, as defined by an anterior-posterior diameter of the spinal canal of <10mm in subjects with lower extremity pain
   3. Neurological deficit possibly associated with the back pain (e.g. foot drop).
   4. Back pain due to pelvic or visceral reasons (e.g.: endometriosis or fibroids) or infection (e.g.: post herpetic neuralgia).
   5. Back pain due to inflammation or damage to the spinal cord or adjacent structures (e.g. arachnoiditis or syringomyelia)
3. Any current indication for back surgery according to local institutional guidelines, or has indication for back surgery but cannot undergo surgery for other reasons.
4. Leg pain described as being worse than back pain, or radiculopathy (neuropathic pain) below the knee.
5. Source of pain is the sacroiliac joint as determined by the Investigator.
6. Drug use
7. Surgical and other procedures exclusions
8. Any prior diagnosis of lumbar vertebral compression fracture, lumbar pars fracture, or lumbar annular tear with disc protrusion
9. Planned surgery.
10. Co-morbid chronic pain conditions
11. Other clinical conditions
12. Psycho-social exclusions
13. Protocol Compliance Exclusions
14. General exclusions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2024-03 (Actual)

PRIMARY OUTCOMES:
11 Point Numerical Rating Scale (NRS) for Low Back Pain | 90 days
Number of subjects with Adverse Events | 90 days, 12 months

SECONDARY OUTCOMES:
Oswestry Disability Index | 90 days

OTHER OUTCOMES:
Subject Global Impression of Change | 90 days

CONTACTS AND LOCATIONS:
Locations (15):
- Australia (5):
  - Pain Medicine of South Australia, Adelaide
  - Hunter Clinical Research, Broadmeadow
  - Metro Spinal Clinic, Caulfield South
  - Precision, Brain, Spine and Pain Centre, Kew
  - Georgius Practice, Noosa
- Belgium (2):
  - GZA Hospitals, Antwerp
  - AZ Nikolaas, Sint-Niklaas
- United Kingdom (8):
  - Basildon & Thurrock University Hospitals, Basildon
  - Southmead Hospital, Bristol
  - Ipswich Hospital, Ipswich
  - Seacroft Hospital, Leeds
  - The Walton Centre, Liverpool
  - St. Bartholomew's Hospital, London
  - James Cook University Hospital, Middlesbrough
  - Southampton University Hospitals, Southampton

REFERENCES:
- [Derived] Thomson S, Williams A, Vajramani G, Sharma M, Love-Jones S, Chawla R, Eldabe S. 5-year longitudinal follow-up of patients treated for chronic mechanical low back pain using restorative neurostimulation. Reg Anesth Pain Med. 2025 Aug 14:rapm-2025-106899. doi: 10.1136/rapm-2025-106899. Online ahead of print. PMID 40813075
- [Derived] Thomson S, Williams A, Vajramani G, Sharma M, Love-Jones S, Chawla R, Eldabe S. Restorative neurostimulation for chronic mechanical low back pain - Three year results from the United Kingdom post market clinical follow-up registry. Br J Pain. 2023 Oct;17(5):447-456. doi: 10.1177/20494637231181498. Epub 2023 Jun 6. PMID 38107760
- [Derived] Thomson S, Chawla R, Love-Jones S, Sharma M, Vajramani G, Williams A, Eldabe S; ReActiv8 PMCF Investigators. Restorative Neurostimulation for Chronic Mechanical Low Back Pain: Results from a Prospective Multi-centre Longitudinal Cohort. Pain Ther. 2021 Dec;10(2):1451-1465. doi: 10.1007/s40122-021-00307-3. Epub 2021 Sep 3. PMID 34478115